CLINICAL TRIAL: NCT04392089
Title: Effects of Cardiovascular and Pulmonary Optimisation on Cerebral Oxygenation in COVID-19 Patients With Severe ARDS
Brief Title: Effects of Cardiovascular and Pulmonary Optimization on Cerebral Oxygenation in COVID-19 Patients With Severe ARDS
Acronym: NIRS-COV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Ana-Marija Hristovska, MD, Ph.d-student, Hvidovre University Hospital
Other Study IDs: H-20027818
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: COVID-19; Respiratory Failure
Keywords: COVID-19; ARDS; NIRS; Saturation
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19: Mechanically ventilated COVID-19 patients with severe ARDS included within 3 days from time of intubation
  Interventions: Device: Masimo, LidCO

INTERVENTIONS:
Device: Masimo, LidCO — * Near-infrared spectroscopy (NIRS), pulse oxymetry (saturation), continous hemoglobine, peripheral perfusion index (PPI) as measured with Massimo
  * Systolic arterial pressure (SAP), diastolic arterial pressure (DAP), mean arterial pressure (MAP), stroke volume (SV), heart rate (HR), cardiac output (CO), systemic vascular resistance (SVR) as measured with LiDCO

SUMMARY:
The aim of the present study is to examine whether cerebral oxygenation could be a more useful parameter than peripheral oxygen saturation to guide clinical titration of permissive hypoxemia in COVID-19 ARDS patients

DETAILED DESCRIPTION:
Mechanical ventilation is the cornerstone of supportive management for most ARDS patients to prevent life-threatening hypoxemia. Arterial oxygenation can be improved via ventilator by increasing fractional inspired oxygen (FiO2) and/or increasing mean airway pressure. When treating mechanically ventilated ARDS patients, the benefit of improved arterial oxygenation must be balanced against the potential risk of ventilator-induced lung injury (VILI), oxygen toxicity occurring with high FiO2 and development of right heart failure.

Arterial oxygen saturation target of 88-95 % and partial oxygen pressure (PaO2) target of 7.3-10.6 are advocated in the management of patients with ARDS. Surprisingly little randomized evidence exists to support these values and current recommendations are thus arbitrary and largely based on normal physiologic values.

Given the lack of evidence of strategies in oxygenating critically ill patients to an oxygen saturation and partial oxygen pressure that is generally accepted to be 'normal,' permissive hypoxemia may offer an alternative that has the potential to improve patient outcomes by avoiding unnecessary harm. Permissive hypoxemia is a concept in which a lower level of arterial oxygenation than usual is accepted in order to avoid the potentially detrimental effects of high fractional inspired oxygen and invasive mechanical ventilation with high pressures, while maintaining adequate oxygen delivery by optimizing cardiac output.

Pulse oximetry is a simple, non-invasive and universally used method to monitor peripheral oxygen saturation of hemoglobin in a variety of clinical settings. Pulse oximetry depends on pulsatile blood flow and only measures the oxyhemoglobin in arterial blood as it leaves the heart. However, this measure does not provide information regarding organ or tissue oxygenation, which reflects the important local balance between oxygen supply and demand.

Near-infrared spectroscopy (NIRS) allows for continuous measurement of regional tissue oxygenation which reflects perfusion status and enables clinicians to directly monitor fluctuations in real time. NIRS reflects the balance of oxygen that is delivered minus what is extracted at tissue level and is an indicator of the tissue oxygen uptake.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Verified COVID-19 infection (throat swab or tracheal aspirate positive for SARS-CoV-2)
* Severe ARDS according to Berlin definition
* Ventilator settings: Controlled IPPV, FiO2 > 0.70, PEEP > 10
* Norepinephrine infusion
* SVV < 10% measured by LiDCO
* RASS - 5

Exclusion Criteria:

* Any of the following contraindications to lung recruitment: pneumothorax, patients on ventilator > 1 week
* Patients with dark pigmented skin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated COVID-19 patients with severe ARDS included within 3 days from time of intubation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in cerebral oxygenation (ScO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization: Step 0 = Baseline, Step 1 = Derecruitment, Step 2 = Recruitment, Step 3 = Norepinephrine challenge, Step 4 = FiO2 increase, Step 5 = FiO2 decrease, Step 6 = Baseline 2

SECONDARY OUTCOMES:
Changes in peripheral oxygen saturation (SatO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in systolic arterial pressure (SAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in diastolic arterial pressure (DAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in mean arterial pressure (MAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in heart rate (HR) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in stroke volume (SV) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in cardiac output (CO) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in systemic vascular resistance (SVR) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in peripheral perfussion index (PPI) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in pH during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in PaO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in PaCO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in arterial saturation (SaO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in PvO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in PvCO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in mixed venous saturation (SvO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in lacatate during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in hemoglobine concentration (Hb) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Changes in muscular oxygenation (SmO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and peripheral oxygen saturation (SatO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and systemic arterial pressure (SAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and diastolic arterial pressure (DAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and mean arterial pressure (MAP) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and stroke volume (SV) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and heart rate (HR) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and cardiac output (CO) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and systemic vascular resistance (SVR) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and peripheral perfussion index (PPI) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and pH during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and PaO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and PaCO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and arterial saturation (SaO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and PvO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and PvCO2 during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and mixed venous saturation (SvO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and lactate during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and hemoglobine concentration (Hb) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above
Association between cerebral oxygenation (ScO2) and muscular oxygenation (SmO2) during cardiovascular and pulmonary optimization | 1 hour
  Cardiovascular and pulmonary optimization as described above

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided